CLINICAL TRIAL: NCT00237380
Title: A Phase 2 Study of PTC124 as an Oral Treatment for Nonsense-Mutation-Mediated Cystic Fibrosis
Brief Title: Safety and Efficacy of Ataluren (PTC124) for Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-005-CF; 20050188
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nonsense mutation; Premature stop codon
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

ARMS (1):
- Ataluren (Experimental): Cycle 1: Within the first 28-day period, ataluren treatment will be taken 3 times per day with meals for 14 days at doses of 4 milligrams/kilogram (mg/kg) (breakfast), 4 mg/kg (lunch), and 8 mg/kg (dinner); there will then be an interval of 14 days without treatment.
  Cycle 2: Within the second 28-day period, ataluren treatment will be taken 3 times per day with meals for 14 days at doses of 10 mg/kg (breakfast), 10 mg/kg (lunch), and 20 mg/kg (dinner); there will then be an interval of 14 days without treatment.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with water.
  Other Names: PTC124

SUMMARY:
In some participants with cystic fibrosis (CF), the disease is caused by a nonsense mutation (premature stop codon) in the gene that makes the cystic fibrosis transmembrane regulator (CFTR) protein. Ataluren has been shown to partially restore CFTR production in animals with CF due to a nonsense mutation. The main purpose of this study is to understand whether ataluren can safely increase functional CFTR protein in the cells of participants with CF due to a nonsense mutation.

DETAILED DESCRIPTION:
In this study, participants with CF due to a nonsense mutation will be treated with a new investigational drug called ataluren. Evaluation procedures to determine if a participant qualifies for the study will be performed within 21 days prior to the start of treatment. Eligible participants who elect to enroll in the study will then participate in two 28-day treatment and follow-up periods (56 days total). There will be a 2-night stay at the clinical research center at the beginning and at the end of each 14 days of ataluren treatment, which means that there will be four 2-night stays at the clinical research center during the study.

One of the measurements for the study is transepithelial potential difference (TEPD), which is also known as nasal potential difference and provides a sensitive evaluation of sodium and chloride transport directly in secretory epithelial cells. TEPD assessments are made on the nasal epithelium cells lining the inferior turbinate because these cells are easier to access than the respiratory epithelial cells lining the lower airways and have been shown to have the same ion transport characteristics. As an endpoint, TEPD has the advantage that it can detect chloride transport changes that are a quantitative integration of the presence, functional activity, and apical location of the CFTR in airway cells. Furthermore, it is a direct measure of CFTR activity that is not likely to be affected by supportive or palliative treatments for CF (with the possible exception of systemically administered aminoglycoside antibiotics).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on documented evidence of a conclusively abnormal sweat test (sweat chloride >60 milliequivalents/litre [mEq/liter]).
* Abnormal chloride secretion as measured by TEPD (a less than -5 mV TEPD assessment of chloride secretion with chloride-free amiloride and isoproterenol).
* Presence of a nonsense mutation in one of the alleles of the CFTR gene.
* Age ≥18 years.
* Body weight ≥40 kg.
* Forced expiratory volume in 1 second (FEV1) ≥40% of predicted for age, gender, and height (Knudson standards).
* Oxygen saturation (as measured by pulse oximetry) ≥92% on room air.
* Willingness of male and female participants, if not surgically sterile, to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and follow-up periods.
* Negative pregnancy test (for females of childbearing potential).
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, and study restrictions.
* Ability to provide written informed consent.

Exclusion Criteria:

* Prior or ongoing medical condition, medical history, physical findings, ECG findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
* Ongoing acute illness including acute upper or lower respiratory infections within 2 weeks before start of study treatment.
* History of major complications of lung disease within 2 months prior to start of study treatment.
* Abnormalities on screening chest x-ray suggesting clinically significant active pulmonary disease other than CF, or new, significant abnormalities that may be indicative of clinically significant active pulmonary involvement secondary to CF.
* Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test.
* Hemoglobin <10 grams per deciliter (g/dL).
* Serum albumin <2.5 g/dL.
* Abnormal liver function (serum alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase [GGT], alkaline phosphatase, lactate dehydrogenase [LDH], or total bilirubin > upper limit of normal).
* Abnormal renal function (serum creatinine >1.5 times upper limit of normal).
* Pregnancy or breast-feeding.
* History of solid organ or hematological transplantation.
* Exposure to another investigational drug within 14 days prior to start of study treatment.
* Ongoing participation in any other therapeutic clinical trial.
* Ongoing use of thiazolidinedione peroxisome proliferator-activated receptor gamma (PPAR γ) agonists, eg, rosiglitazone (Avandia® or equivalent) or pioglitazone (Actos® or equivalent)
* Change in intranasal medications (including use of corticosteroids, cromolyn, ipratropium bromide, phenylephrine, or oxymetazoline) within 14 days prior to start of study treatment.
* Change in treatment with systemic or inhaled corticosteroids within 14 days prior to start of study treatment.
* Use or requirement for inhaled gentamicin or amikacin within 14 days prior to start of study treatment or during study treatment.
* Requirement for systemic aminoglycoside antibiotics within 14 days prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-11-30 (Actual); Primary Completion 2006-05-31 (Actual); Study Completion 2006-05-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to End of Treatment in Total Chloride Transport | Baseline of Cycle 1 and Cycle 2, Day 14 and Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Number of Participants With a Chloride Transport Response | Baseline of Cycle 1 and Cycle 2 and Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Number of Participants With a Chloride Transport Normalization Between Baseline and End of Treatment | Baseline of Cycle 1 and Cycle 2 and Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)

SECONDARY OUTCOMES:
Change From Baseline in Nasal Chloride Secretion as Assessed by Transepithelial Potential Difference (TEPD) | Baseline of Cycle 1 and Cycle 2, Day 14 and Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Change From Baseline in Sweat Chloride Concentration as Determined by Pilocarpine Iontophoresis | Baseline, Day 41
Change From Baseline in CFTR Protein in Nasal Mucosa as Determined by Immunofluorescence | Baseline of Cycle 1 and Cycle 2, Day 14 and Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Change From Baseline in Nonsense Mutation CFTR mRNA in Nasal Mucosa as Determined by Quantitative Polymerase Chain Reaction (PCR) Assay | Baseline of Cycle 1 and Cycle 2, Day 14 and Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Change From Baseline in Number of Neutrophils in Blood | Baseline Up to Day 56
Change From Baseline in Pulmonary Function as Measured by Spirometry | Baseline of Cycle 1 and Cycle 2, Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Change From Baseline in Body Weight | Baseline of Cycle 1 and Cycle 2, Day 28 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Compliance with Study Treatment | Baseline Up to Day 56
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of Ataluren | 0 (predose), 1, 2, 3, and 4 hours (hrs) postdose of the midday dose; 0 (predose), 1, 2, 3, 4, and 12 hrs postdose of the evening dose on Day 1 and Day 27
PK: Maximum Plasma Concentration (Cmax) of Ataluren | 0 (predose), 1, 2, 3, and 4 hrs postdose of the morning dose; 0 (predose), 1, 2, 3, and 4 hrs postdose of the midday dose; and 0 hrs (predose), 1, 2, 3, 4, and 12 hrs postdose of the evening dose on Days 1 and 13 of Cycles 1 and 2 (1 cycle=28 days)
PK: Area Under the Plasma Concentration Time Curve (AUC) of Ataluren | 0 (predose), 1, 2, 3, and 4 hrs postdose of the morning dose; 0 (predose), 1, 2, 3, and 4 hrs postdose of the midday dose; and 0 hrs (predose), 1, 2, 3, 4, and 12 hrs postdose of the evening dose on Days 1 and 13 of Cycles 1 and 2 (1 cycle=28 days)
PK: Terminal Elimination Half Life (T1/2) of Ataluren | 0 (predose), 1, 2, 3, and 4 hrs postdose of the morning dose; 0 (predose), 1, 2, 3, and 4 hrs postdose of the midday dose; and 0 hrs (predose), 1, 2, 3, 4, and 12 hrs postdose of the evening dose on Days 1 and 13 of Cycles 1 and 2 (1 cycle=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Eiten Kerem, MD, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital - Mount Scopus, Jerusalem, Israel

REFERENCES:
- [Derived] Kerem E, Hirawat S, Armoni S, Yaakov Y, Shoseyov D, Cohen M, Nissim-Rafinia M, Blau H, Rivlin J, Aviram M, Elfring GL, Northcutt VJ, Miller LL, Kerem B, Wilschanski M. Effectiveness of PTC124 treatment of cystic fibrosis caused by nonsense mutations: a prospective phase II trial. Lancet. 2008 Aug 30;372(9640):719-27. doi: 10.1016/S0140-6736(08)61168-X. Epub 2008 Aug 20. PMID 18722008